CLINICAL TRIAL: NCT02482675
Title: Regulation of Postprandial Nitric Oxide Bioavailability and Vascular Function By Dairy Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor and Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015H0088
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Prediabetes
Keywords: Dairy; Milk; Glucose; Postprandial; Hyperglycemia; Prediabetes; Blood glucose; Oxidative stress; Vascular health; Vascular function
MeSH Terms: conditions — Prediabetic State; Hyperglycemia | interventions — Glucose; Caseins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glucose (Active Comparator): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose
- Glucose with Non-fat Milk (Experimental): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose with Non-fat Milk
- Glucose with Whey Protein Isolate (Experimental): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose with Whey Protein Isolate
- Glucose with Sodium Caseinate (Experimental): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose with Sodium Caseinate

INTERVENTIONS:
Other: Glucose — Following baseline measurements, participants will consume a 75 g glucose solution within five minutes.
  Arms: Glucose
Other: Glucose with Non-fat Milk — Following baseline measurements, participants will consume 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Arms: Glucose with Non-fat Milk
Other: Glucose with Whey Protein Isolate — Following baseline measurements, participants will consume 75 g glucose and whey protein isolate dissolved in 2 cups water within five minutes.
  Arms: Glucose with Whey Protein Isolate
Other: Glucose with Sodium Caseinate — Following baseline measurements, participants will consume 75 g glucose and sodium caseinate dissolved in 2 cups water within five minutes.
  Arms: Glucose with Sodium Caseinate

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Short-term increases in blood sugar, or postprandial hyperglycemia (PPH), affect blood vessel function and increase the risk of CVD. Greater intakes of dairy foods have been associated with a lower risk of CVD, but whether these effects occur directly or indirectly by displacing foods in the diet that might increase CVD risk is unclear. The health benefits of dairy on heart health are at least partly attributed to its ability to limit PPH and resulting PPH-mediated responses leading to vascular dysfunction. This provides rationale to further investigate dairy as a dietary strategy to reduce PPH and risk for CVD. The objective of this study is to define the extent to which dairy milk, and its whey and casein protein fractions, protect against postprandial vascular dysfunction by reducing oxidative stress responses that limit nitric oxide bioavailability to the vascular endothelium in adults with prediabetes.

DETAILED DESCRIPTION:
This study consists of four, 3-hour postprandial trials in response to consuming the following dietary treatments: 1. oral glucose challenge, 2. oral glucose challenge in combination with non-fat milk, 3. oral glucose challenge in combination with whey protein isolate, and 4. oral glucose challenge in combination with sodium caseinate. For three days preceding each trial, participants will be provided all meals to standardize physiologic responses to test meals. On each trial day, vascular function will be assessed and blood samples collected prior to and at 30 minute intervals for 3 hours following test meal ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. hemoglobin A1c 5.7-6.4%
2. non-dietary supplement user
3. no medications affecting vasodilation, inflammation, or energy metabolism
4. no CVD
5. nonsmokers
6. individuals having blood pressure <140/90 mmHg and total cholesterol <240 mg/dL

Exclusion Criteria:

1. unstable weight (±2 kg)
2. vegetarian or dairy allergy
3. alcohol intake >3 drinks/day or >10 drinks/week
4. ≥7 hours/week of aerobic activity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] DECODE Study Group, the European Diabetes Epidemiology Group.. Glucose tolerance and cardiovascular mortality: comparison of fasting and 2-hour diagnostic criteria. Arch Intern Med. 2001 Feb 12;161(3):397-405. doi: 10.1001/archinte.161.3.397. PMID 11176766
- [Background] Ballard KD, Bruno RS. Protective role of dairy and its constituents on vascular function independent of blood pressure-lowering activities. Nutr Rev. 2015 Jan;73(1):36-50. doi: 10.1093/nutrit/nuu013. PMID 26024056
- [Background] Ballard KD, Mah E, Guo Y, Pei R, Volek JS, Bruno RS. Low-fat milk ingestion prevents postprandial hyperglycemia-mediated impairments in vascular endothelial function in obese individuals with metabolic syndrome. J Nutr. 2013 Oct;143(10):1602-10. doi: 10.3945/jn.113.179465. Epub 2013 Aug 21. PMID 23966328
- [Background] McDonald JD, Mah E, Chitchumroonchokchai C, Dey P, Labyk AN, Villamena FA, Volek JS, Bruno RS. Dairy milk proteins attenuate hyperglycemia-induced impairments in vascular endothelial function in adults with prediabetes by limiting increases in glycemia and oxidative stress that reduce nitric oxide bioavailability. J Nutr Biochem. 2019 Jan;63:165-176. doi: 10.1016/j.jnutbio.2018.09.018. Epub 2018 Sep 25. PMID 30412905

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucose, Then Whey Protein, Then Sodium Caseinate, Then Milk; Glucose, Then Milk, Then Sodium Caseinate, Then Whey Protein; Glucose, Then Sodium Caseinate, Then Milk, Then Whey Protein; Glucose, Then Whey Protein, Then Milk, Then Sodium Caseinate; Glucose, Then Sodium Caseinate, Then Whey Protein, Then Milk; Milk, Then Glucose, Then Sodium Caseinate, Then Whey Protein; Milk, Then Whey Protein, Then Glucose, Then Sodium Caseinate; Milk, Then Whey Protein, Then Sodium Caseinate, Then Glucose; Milk, Then Sodium Caseinate, Then Whey Protein, Then Glucose; Milk, Then Glucose, Then Whey Protein, Then Sodium Caseinate; Milk, Then Sodium Caseinate, Then Glucose, Then Whey Protein; Whey Protein, Then Glucose, Then Sodium Caseinate, Then Milk; Whey Protein, Then Glucose, Then Milk, Then Sodium Caseinate; Whey Protein, Then Sodium Caseinate, Then Glucose, Then Milk; Whey Protein, Then Milk, Then Sodium Caseinate, Then Glucose; Whey Protein, Then Sodium Caseinate, Then Milk, Then Glucose; Whey Protein, Then Milk, Then Glucose, Then Sodium Caseinate; Sodium Caseinate, Then Glucose, Then Milk, Then Whey Protein; Sodium Caseinate, Then Whey Protein, Then Milk, Then Glucose; Sodium Caseinate, Then Milk, Then Glucose, Then Whey Protein; Sodium Caseinate, Then Whey Protein, Then Glucose, Then Milk; Sodium Caseinate, Then Milk, Then Whey Protein, Then Glucose; Sodium Caseinate, Then Glucose, Then Whey Protein, Then Milk: Each study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Glucose: Following baseline measurements, participants will consume a 75 g glucose solution within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants will consume 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose with Whey Protein Isolate: Following baseline measurements, participants will consume 75 g glucose and whey protein isolate dissolved in 2 cups water within five minutes.
  Glucose with Sodium Caseinate: Following baseline measurements, participants will consume 75 g glucose and sodium caseinate dissolved in 2 cups water within five minutes.
Period: Overall Study
Arm/Group | Glucose, Then Whey Protein, Then Sodium Caseinate, Then Milk | Glucose, Then Milk, Then Sodium Caseinate, Then Whey Protein | Glucose, Then Sodium Caseinate, Then Milk, Then Whey Protein | Glucose, Then Whey Protein, Then Milk, Then Sodium Caseinate | Glucose, Then Sodium Caseinate, Then Whey Protein, Then Milk | Milk, Then Glucose, Then Sodium Caseinate, Then Whey Protein | Milk, Then Whey Protein, Then Glucose, Then Sodium Caseinate | Milk, Then Whey Protein, Then Sodium Caseinate, Then Glucose | Milk, Then Sodium Caseinate, Then Whey Protein, Then Glucose | Milk, Then Glucose, Then Whey Protein, Then Sodium Caseinate | Milk, Then Sodium Caseinate, Then Glucose, Then Whey Protein | Whey Protein, Then Glucose, Then Sodium Caseinate, Then Milk | Whey Protein, Then Glucose, Then Milk, Then Sodium Caseinate | Whey Protein, Then Sodium Caseinate, Then Glucose, Then Milk | Whey Protein, Then Milk, Then Sodium Caseinate, Then Glucose | Whey Protein, Then Sodium Caseinate, Then Milk, Then Glucose | Whey Protein, Then Milk, Then Glucose, Then Sodium Caseinate | Sodium Caseinate, Then Glucose, Then Milk, Then Whey Protein | Sodium Caseinate, Then Whey Protein, Then Milk, Then Glucose | Sodium Caseinate, Then Milk, Then Glucose, Then Whey Protein | Sodium Caseinate, Then Whey Protein, Then Glucose, Then Milk | Sodium Caseinate, Then Milk, Then Whey Protein, Then Glucose | Sodium Caseinate, Then Glucose, Then Whey Protein, Then Milk
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Glucose: Following baseline measurements, participants will consume a 75 g glucose solution within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants will consume 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose with Whey Protein Isolate: Following baseline measurements, participants will consume 75 g glucose and whey protein isolate dissolved in 2 cups water within five minutes.
  Glucose with Sodium Caseinate: Following baseline measurements, participants will consume 75 g glucose and sodium caseinate dissolved in 2 cups water within five minutes.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (4.3)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 106.9 (14.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125.3 (9.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 83 (7.5)
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.8 (0.4)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.6 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Vascular Endothelial Function
Description: Flow mediated dilation (FMD) of the brachial artery, calculated as FMD AUC for 0-180 minutes (change from baseline)
Time Frame: Area under curve for FMD for three hours (0, 30, 60, 90, 120, 180 minutes)
Measure: Mean (Standard Error); unit: %*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
%*min | -307 (67.1) | -34.8 (62) | -36.8 (63.3) | -110 (49.8)

2. Secondary Outcome: Nitrite/Nitrate (NOx)
Description: NOx AUC for 0-180 minutes
Time Frame: Area under curve for nitrite/nitrate for three hours (0, 30, 60, 90, 120, 180 min) (change from baseline)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
umol/L*min | -1363 (285) | 347 (329) | -21 (207) | -57.2 (237)

3. Secondary Outcome: Plasma Glucose
Description: Plasma glucose concentration from 0-180 minutes
Time Frame: Area under the curve for glucose for three hours (0, 30, 60, 90, 120, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: mg/dL*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
mg/dL*min | 5828 (669) | 4032 (702) | 3340 (619) | 3640 (550)

4. Secondary Outcome: Malondialdehyde (MDA)
Description: Plasma MDA measured as MDA AUC from 0-180 minutes
Time Frame: Area under curve for MDA for three hours (0, 30, 60, 90, 120, 150, 180 min.) (change from baseline)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
umol/L*min | 66.5 (6.06) | 43.2 (4.27) | 46.4 (4.34) | 45.1 (3.56)

5. Secondary Outcome: Arginine (ARG)
Description: Plasma arginine concentration, calculated as ARG AUC from 0-180 minutes
Time Frame: ARG area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
umol/L*min | -3922 (486) | -1235 (565) | 195 (632) | -189 (628)

6. Secondary Outcome: Asymmetric Dimethylarginine/Arginine (ADMA/ARG)
Description: Plasma ADMA/arginine concentration, calculated as ADMA/ARG AUC from 0-180 minutes
Time Frame: ADMA/ARG area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: (nmol/L)/(umol/L)*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
(nmol/L)/(umol/L)*min | 275 (34) | 55 (43) | 47 (38) | 25 (37)

7. Secondary Outcome: Symmetric Dimethylarginine/Arginine (SDMA/ARG)
Description: Plasma SDMA/arginine concentration, calculated as SDMA/ARG AUC from 0-180 minutes
Time Frame: SDMA/ARG area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: (nmol/L)/(umol/L)*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
(nmol/L)/(umol/L)*min | 175 (14) | 31 (13) | 4 (16) | -17 (12)

8. Secondary Outcome: Tetrahydrobiopterin/Dihydrobiopterin (BH4/BH2)
Description: Plasma BH4/BH2 concentration, calculated as BH4/BH2 AUC from 0-180 minutes
Time Frame: Plasma BH4/BH2 concentration area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: ratio*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
ratio*min | -47 (119) | 78 (99) | 171 (122) | 131 (67)

9. Secondary Outcome: Insulin
Description: Plasma insulin concentration, calculated as insulin AUC from 0-180 minutes
Time Frame: Insulin area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: uIU/mL*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
uIU/mL*min | 8179.7 (904.91) | 8196.1 (882.03) | 8654.6 (804.32) | 8656.9 (869.98)

10. Secondary Outcome: Cholecystokinin (CCK)
Description: Plasma CCK concentration, calculated as CCK AUC from 0-180 minutes
Time Frame: CCK area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: pmol/L*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
pmol/L*min | 89.67 (117.52) | 422.87 (182.43) | 352.5 (154.03) | 519.94 (202.36)

11. Secondary Outcome: 8-isoprostaglandin-F2a
Description: Plasma 8-isoprostaglandin-F2a concentration, calculated as 8-isoprostaglandin-F2a AUC from 0-180 minutes
Time Frame: 8-isoprostaglandin-F2a area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: pg/mL*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
pg/mL*min | 2162.2 (436.50) | -824.14 (368.68) | -18.75 (498.80) | 229.14 (484.62)

12. Secondary Outcome: 8-isoprostaglandin-F2a/Arachidonic Acid
Description: Plasma 8-isoprostaglandin-F2a/Arachidonic acid concentration, calculated as 8-isoprostaglandin-F2a/Arachidonic acid AUC from 0-180 minutes
Time Frame: 8-isoprostaglandin-F2a/Arachidonic acid area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: (pg/mL)/(ug/mL)*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
(pg/mL)/(ug/mL)*min | 10129 (1613.7) | -1655.2 (1477.1) | 2422.3 (2030.6) | 3907.6 (2378.7)

13. Secondary Outcome: Arachidonic Acid
Description: Arachidonic acid concentration, calculated as Arachidonic acid AUC from 0-180 minutes
Time Frame: Arachidonic acid area under the curve for 3 hours (0, 30, 60, 90, 120, 150, 180 minutes) (change from baseline)
Measure: Mean (Standard Error); unit: ug/mL*min
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Number analyzed (Participants) | 23 | 23 | 23 | 23
ug/mL*min | -2570 (451.86) | -1358.4 (497.54) | -2762.6 (529.07) | -2752.0 (462.74)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during the entirety of the study duration (~6 total weeks).
Description: Participants completed a cross-over trial that examined blood vessel function and related biomarkers in response to a single controlled meal.
Arm/Group | Glucose | Glucose With Non-fat Milk | Glucose With Whey Protein Isolate | Glucose With Sodium Caseinate
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No